CLINICAL TRIAL: NCT00904748
Title: A Relative Bioavailability Study Between Two Formulations Of Sildenafil Citrate In Healthy Male Subjects, Fasting Dosing, Being The Test Formulation Sildenafil Citrate 100 Mg CT , And The Reference Formulation Sildenafil Citrate 100 Mg Film-Coated Tablets (Viagra®), Both Formulations Manufactured By Laboratórios Pfizer Ltda.
Brief Title: A Relative Bioavailability Study Between Two Formulations Of Sildenafil Citrate
Acronym: A1481272
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A1481272; JPJ 39/09
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2011-04-04 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: Sildenafil; Bio-equivalence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test 1 (Experimental)
  Interventions: Drug: sildenafil citrate 100 mg CT
- Test 2 (Experimental)
  Interventions: Drug: sildenafil citrate 100 mg CT
- Reference (Active Comparator)
  Interventions: Drug: Viagra®

INTERVENTIONS:
Drug: sildenafil citrate 100 mg CT — sildenafil citrate 100 mg CT, single dose without water
  Arms: Test 1
Drug: sildenafil citrate 100 mg CT — sildenafil citrate 100 mg CT, single dose with water
  Arms: Test 2
Drug: Viagra® — sildenafil citrate 100 mg film-coated tablet (Viagra®), single dose
  Arms: Reference

SUMMARY:
The purpose of this study is to perform a relative bioavailability study between two formulations of sildenafil citrate.

DETAILED DESCRIPTION:
Bio-equivalence between two formulations of sildenafil citrate

ELIGIBILITY:
Inclusion Criteria:

* Body mass index higher or equal to 18,5 and lower or equal than 29,9 kg/m2.
* Good health conditions or without significant disease, at medical discretion, according to the rules defined in the Protocol, and evaluations undergone: clinical history, pulse and blood pressure measurements, physical and psychological examination, ECG and complementary laboratory examination.
* Able to understand the study nature and objective, including the risks and adverse effects and willing to cooperate with the investigator and act according to all the trial requirements, which is confirmed by signing the Informed Consent Form.

Exclusion Criteria:

* Hypersensitivity to the study drug or to the chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug.
* History or presence of hepatic or gastrointestinal diseases, or other condition that affects the drug absorption, distribution, excretion or metabolism
* History of hepatic, renal, lung, gastrointestinal, epileptic, hematological or psychiatric disease; hypo or hypertension of whatever etiology which demands treatment with drugs; history or occurrence of myocardial infarction, angina and/or cardiac failure;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Bragança Paulista, São Paulo, Brazil

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481272&StudyName=A%20Relative%20Bioavailability%20Study%20Between%20Two%20Formulations%20Of%20Sildenafil%20Citrate

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant was to receive each of 3 formulations in 3 treatment periods, after being allocated to 1 of 6 treatment sequences. There was to be a minimum interval of 3 days between treatment periods.
Groups:
- Sequence 1: Reference (Sildenafil 100 milligram (mg) coated tablet administered with water, Test 1 (Sildenafil 100 milligram (mg) chewable tablet administered without water), Test 2 (Sildenafil 100 milligram (mg) chewable tablet administered with water)
- Sequence 2: Reference (Sildenafil 100 milligram (mg) coated tablet administered with water, Test 2 (Sildenafil 100 milligram (mg) chewable tablet administered with water), Test 1 (Sildenafil 100 milligram (mg) chewable tablet administered without water)
- Sequence 3: Test 1 (Sildenafil 100 milligram (mg) chewable tablet administered without water), Reference (Sildenafil 100 milligram (mg) coated tablet administered with water, Test 2 (Sildenafil 100 milligram (mg) chewable tablet administered with water)
- Sequence 4: Test 1 (Sildenafil 100 milligram (mg) chewable tablet administered without water), Test 2 (Sildenafil 100 milligram (mg) chewable tablet administered with water), Reference (Sildenafil 100 milligram (mg) coated tablet administered with water
- Sequence 5: Test 2 (Sildenafil 100 milligram (mg) chewable tablet administered with water), Reference (Sildenafil 100 milligram (mg) coated tablet administered with water, Test 1 (Sildenafil 100 milligram (mg) chewable tablet administered without water)
- Sequence 6: Test 2 (Sildenafil 100 milligram (mg) chewable tablet administered with water), Test 1 (Sildenafil 100 milligram (mg) chewable tablet administered without water), Reference (Sildenafil 100 milligram (mg) coated tablet administered with water
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 (1 participant randomized to this sequence discontinued prior to receipt of study medication.) | 8
Received Treatment | 8 | 8 | 8 | 8 | 7 | 8
Completed | 7 | 7 | 7 | 6 | 7 | 8
Not Completed | 1 | 1 | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants who were randomized to any treatment sequence
Arm/Group | Entire Study Population
Number analyzed (Participants) | 48
Age, Continuous [Mean (Full Range); unit: years] | 29.3 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC 0-t)
Description: Area under the blood concentration-time profile from time zero to last experimentally determined concentration measured in nanograms*hour/milliliter (ng*hr/mL).
Time Frame: Day 1 (Period 1), Day 8 (Period 2), and Day 15 (Period 3): Pre-dose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours post-dose
Population: Participants for pharmacokinetic analysis = participants who completed all of the 3 treatment periods.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Test 1: 100 mg Chewable, Without Water: Test 1 Formulation: Sildenafil citrate 100 milligram (mg) chewable tablet administered without water
- Test 2: 100 mg Chewable, With Water: Test 2 Formulation: Sildenafil citrate 100 mg chewable tablet administered with water
- Reference: 100 mg Coated, With Water: Reference Formulation: Viagra (sildenafil citrate) 100 mg coated tablet administered with water
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water
Number analyzed (Participants) | 42 | 42 | 42
ng*hr/mL | 1467.00 (560.99) | 1458.45 (602.73) | 1493.53 (615.59)
Statistical Analysis 1: Comparison: Test 1: 100 mg Chewable, Without Water vs Reference: 100 mg Coated, With Water; Ratio between geometric means of Test 1 study treatment (chewable without water) and reference study treatment (coated with water); Test type: Non-Inferiority or Equivalence — Percent of reference to detect for 2-1 tests and power = 20.0%; ANOVA; ratio between geometric means = 98.68, 90% CI 2-sided [92.03 to 105.82] — Estimated value = ratio (% reference)
Statistical Analysis 2: Comparison: Test 2: 100 mg Chewable, With Water vs Reference: 100 mg Coated, With Water; Ratio between geometric means of Test 2 study treatment (chewable with water) and reference study treatment (coated with water); Test type: Non-Inferiority or Equivalence — Percent of reference to detect for 2-1 tests and power = 20.0%; ANOVA; ratio between geometric means = 97.23, 90% CI 2-sided [90.67 to 104.26] — Estimated value = ratio (% reference)

2. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration measured in nanograms per milliliter (ng/mL).
Time Frame: as for outcome 1
Population: Participants for pharmacokinetic analysis = participants who completed all of the 3 treatment periods.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water
Number analyzed (Participants) | 42 | 42 | 42
ng/mL | 439.38 (198.25) | 434.38 (211.53) | 532.31 (217.32)
Statistical Analysis 1: Comparison: Test 1: 100 mg Chewable, Without Water vs Reference: 100 mg Coated, With Water; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Percent of reference to detect for 2-1 tests and power = 20%; ANOVA; ratio between geometric means = 80.83, 90% CI 2-sided [72.38 to 90.26] — Estimated value = ratio (% reference)
Statistical Analysis 2: Comparison: Test 2: 100 mg Chewable, With Water vs Reference: 100 mg Coated, With Water; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — Percent of reference to detect for 2-1 tests and power = 20%; ANOVA; ratio between geometric means = 78.76, 90% CI 2-sided [70.53 to 87.96] — Estimated value = ratio (% reference)

3. Secondary Outcome: Area Under the Curve From 0 to Infinity (AUC 0-inf )
Description: Area under the blood concentration-time profile from time zero extrapolated to infinite time measured in nanograms *hour/milliliter (ng*hr/mL).
Time Frame: as for outcome 1
Population: Participants for pharmacokinetic analysis = participants who completed all of the 3 treatment periods.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water
Number analyzed (Participants) | 42 | 42 | 42
ng*hr/mL | 1547.92 (588.48) | 1534.66 (618.86) | 1573.81 (648.32)
Statistical Analysis 1: Comparison: Test 1: 100 mg Chewable, Without Water vs Reference: 100 mg Coated, With Water; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Percent of reference to detect for 2-1 tests and power = 20.0%; ANOVA; ratio between geometric means = 99.12, 90% CI 2-sided [92.76 to 105.93] — Estimated value = ratio (% reference)
Statistical Analysis 2: Comparison: Test 2: 100 mg Chewable, With Water vs Reference: 100 mg Coated, With Water; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — Percent of reference to detect for 2-1 tests and power = 20.0%; ANOVA; ratio between geometric means = 97.84, 90% CI 2-sided [91.56 to 104.56] — Estimated value = ratio (% reference)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time at which maximum plasma concentration (Cmax) occurred.
Time Frame: as for outcome 1
Population: Participants for pharmacokinetic analysis = participants who completed all of the 3 treatment periods.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water
Number analyzed (Participants) | 42 | 42 | 42
hours | 1.46 (0.81) | 1.29 (0.71) | 1.28 (0.85)
Statistical Analysis 1: Comparison: Test 1: 100 mg Chewable, Without Water vs Reference: 100 mg Coated, With Water; Difference in Tmax between Test 1 study treatment (chewable without water) and reference study treatment (coated with water); Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.18, 90% CI 2-sided [-0.14 to 0.50]
Statistical Analysis 2: Comparison: Test 2: 100 mg Chewable, With Water vs Reference: 100 mg Coated, With Water; Difference in Tmax between Test 2 study treatment (chewable with water) and reference study treatment (coated with water); Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.27 to 0.28]

5. Secondary Outcome: Half-life (T 1/2)
Description: Terminal elimination half-life.
Time Frame: as for outcome 1
Population: Participants for pharmacokinetic analysis = participants who completed all of the 3 treatment periods.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water
Number analyzed (Participants) | 42 | 42 | 42
hours | 2.96 (0.63) | 2.84 (0.74) | 2.93 (0.81)

6. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Clinically significant abnormalities in blood pressure (BP), pulse, and temperature reported as an adverse event. Clinically significant = values outside the normal range and/or values judged as significant by the investigator (normal range: systolic BP 100-140 mmHg; diastolic BP 60- 90 mmHg; temperature 35-37°Celsius). Pulse rate based on investigator discretion.
Time Frame: Day 1 (Period 1), Day 8 (Period 2), and Day 15 (Period 3): Pre-dose and 0.5, 1, 2, 4, 8 and 12 hours post-dose.
Population: Safety population: all subjects who received at least 1 dose of study medication. Although individual listing data for vital signs were collected, summary statistics were not generated for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water
Number analyzed (Participants) | 47 | 47 | 47
participants | 0 | 1 | 0

ADVERSE EVENTS:
Description: Safety population: subjects who received at least 1 dose of study medication in any treatment period. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and non-serious for another subject or subject may have had a serious and non-serious episode of same event.
Groups:
- Formulation Unspecified: Sildenafil 100 mg tablet: formulation unspecified
Arm/Group | Test 1: 100 mg Chewable, Without Water | Test 2: 100 mg Chewable, With Water | Reference: 100 mg Coated, With Water | Formulation Unspecified
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 3/47 | 3/47 | 3/47 | 18/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test 1: 100 mg Chewable, Without Water (N=47) | Test 2: 100 mg Chewable, With Water (N=47) | Reference: 100 mg Coated, With Water (N=47) | Formulation Unspecified (N=47)
Headache (General disorders) | 3 | 2 | 2 | 0
Nausea (General disorders) | 1 | 0 | 1 | 0
Loose stools (General disorders) | 1 | 0 | 0 | 0
Hypotension (General disorders) | 0 | 1 | 0 | 0
Vomiting (General disorders) | 0 | 0 | 1 | 0
Laboratory change: urine (General disorders) | 0 | 0 | 0 | 8
Laboratory change: red blood cell count (General disorders) | 0 | 0 | 0 | 4
Laboratory change: triglycerides (General disorders) | 0 | 0 | 0 | 2
Laboratory change: glucose (General disorders) | 0 | 0 | 0 | 3
Laboratory change: cholesterol (General disorders) | 0 | 0 | 0 | 2
Laboratory change: white blood cells (General disorders) | 0 | 0 | 0 | 1
Laboratory changes unspecified (General disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.